CLINICAL TRIAL: NCT07295730
Title: Use of 3D-printed Models and Augmented Reality in Medical Student Education of Congenital Heart Disease: Randomized Controlled Trial
Brief Title: 3D Modalities for Medical Student Education of Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY20240627
Record Dates: First submitted 2025-12-10; First posted 2025-12-22 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Tetralogy of Fallot (TOF); Hypoplastic Left Heart Syndrome (HLHS)
MeSH Terms: conditions — Tetralogy of Fallot; Hypoplastic Left Heart Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Slide-based lecture (Other): Participants in this group received teaching using a slide-based lecture
  Interventions: Other: 3D-printed heart models and augmented reality
- 3D-printed Model (Active Comparator): This group received teaching using 3D-printed models
  Interventions: Other: 3D-printed heart models and augmented reality
- Augmented Reality (Active Comparator): This group received teaching using augmented reality headsets
  Interventions: Other: 3D-printed heart models and augmented reality

INTERVENTIONS:
Other: 3D-printed heart models and augmented reality — Participants will receive an educational session regarding congenital heart disease using a slide-based lecture, 3D-printed models, or augmented reality headsets.

SUMMARY:
The goal of this clinical trial is to learn if 3D-printed heart models and augmented reality can be useful modalities to teach medical students about congenital heart disease. The main questions it aims to answer are:

1. Does using 3D-printed heart models improve learners' understanding of congenital heart disease when compared to traditional slide-based teaching methods?
2. Does using augmented reality heart models improve learners' understanding of congenital heart disease when compared to traditional slide-based teaching methods?
3. How can these modalities best be integrated into standard medical school curricula?

Participants will:

1. Take a pre-test consisting of questions regarding anatomy and physiology of the normal heart as well as two congenital heart diseases.
2. Be randomized into 3 groups that receive a teaching session using either slide-based lecture, 3D-printed models, or augmented reality.
3. Take a post-test of the same questions from the pre-test.
4. Take a delayed post-test of the same questions with additional subjective questions about their experience with their assigned modality.

ELIGIBILITY:
Inclusion Criteria:

* First year medical student

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2025-11-20 (Actual); Primary Completion 2025-12-09 (Actual); Study Completion 2025-12-09 (Actual)

PRIMARY OUTCOMES:
Changes in Pre and Post-test Scores | Enrollment Pre-Intervention, Baseline Post-Intervention, and 3 Weeks Post-Intervention
  Participants completed a 16-item, multiple choice questionnaire about the anatomy and physiology of the normal heart and two complex congenital heart defects. The questionnaire is broken down into 4 questions on basic cardiology and 6 questions each pertaining specifically to tetralogy of Fallot and hypoplastic left heart syndrome. The questionnaire is delivered pre-intervention, immediately post-intervention, and again at 3-weeks post intervention. Correct answers are scored as true (1) and incorrect answers scored as false (0) with a score range of 0-16 with higher scores indicating better retention and understanding of the curriculum.

CONTACTS AND LOCATIONS:
Overall Officials: Arpit Agarwal, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Case Western Reserve University School of Medicine, Cleveland, Ohio, United States

DOCUMENTS (1):
  • Study Protocol (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/30/NCT07295730/Prot_000.pdf